CLINICAL TRIAL: NCT03614351
Title: The Effects of Providing Protein and Nutritional Guidance on Healing Times After ACL Surgery
Brief Title: Dietary Protein Intake and Rehabilitation From Anterior Cruciate Ligament Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding to pay for a coordinator and interventionist,
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00046590
Record Dates: First submitted 2018-07-25; First posted 2018-08-03 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2020-07

CONDITIONS: ACL Injury
Keywords: protein; nutritional guidance; ACL surgery
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Proteins

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Physical therapy staff will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Therapy plus Protein Supplement (Experimental): Participants will be randomized to the protein supplementation group, PROT, and will receive education from a dietary counselor on how to monitor protein intake using a smartphone app.
  Interventions: Dietary Supplement: Protein (PROT)
- Physical Therapy Control (Active Comparator): Participants will be randomized to the enhanced-care control group, CONT, and will receive education from a dietary counselor on how to monitor protein intake using a smartphone app.
  Interventions: Other: Control (CONT)

INTERVENTIONS:
Dietary Supplement: Protein (PROT) — Participants will receive Combat Protein Powder made by MusclePharm in an amount sufficient to take 80g daily until their next visit. They will be encouraged to ingest 40 g after exercise and 40 g before bed which will partly comprise their daily goal. They will be educated on the concept of complete high quality proteins, and that some proteins can facilitate muscle growth greater than others. Additionally, they will receive meal plan ideas and shopping tips that will facilitate healthy and economical protein consumption up to or beyond their daily goal.
  Arms: Physical Therapy plus Protein Supplement
Other: Control (CONT) — Instructed not to alter their diet based on the app, and to continue to eat as they normally would.
  Arms: Physical Therapy Control

SUMMARY:
Protein supplementation may promote increases in strength and hypertrophy in the context of resistance training (RT) and reduce markers of inflammation, while sufficient levels of protein are necessary for healing certain wounds and maintenance of muscle mass in a protein depleted state. Protein supplementation could be useful to improve clinical outcomes.

DETAILED DESCRIPTION:
Protein supplementation may promote increases in strength and hypertrophy in the context of resistance training (RT) and reduce markers of inflammation, while sufficient levels of protein are necessary for healing certain wounds and maintenance of muscle mass in a protein depleted state. Despite this, no studies have investigated the role of protein provision in the context of physical therapy (PT) or musculoskeletal rehabilitation, including following surgical interventions. Survey data of Americans in the highest protein consuming age range (19-30 year old consuming 91 g/kg body weight/day), show they have an adequate protein intake to maintain nitrogen balance at baseline (85 g/kg). However, if patients under consume protein, as apparent in older adults (mean intake of 66 g/kg) these individuals will require more during times of tissue healing or could benefit with more in attempting to build back their strength through RT or PT. Thus, protein supplementation could be useful to improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a complete ACL tear and received a hamstring autograft ACL repair surgery (within 8 months of injury) and plan to complete physical therapy and follow up treatment with WFBH at D1 outpatient rehabilitation
* Subjects must have a smartphone capable of running the nutrition tracking app (My Fitness Pal)

Exclusion Criteria:

* Subjects must not have other ligamentous involvement, or complications during the surgical procedure.
* They must not have had a concurrent meniscal repair (debridement is acceptable).
* They must not have post-operative limitations that interfere with rehabilitation.
* Patients determined by the referring surgeon to be poor candidates for the study for any medical (including history of eating disorder, phenylketonuria, maple syrup urine disease, food allergies, lactose intolerance, kidney or liver disease) or other reasons that deem them inappropriate to complete the intervention (driving distance from facility, work schedule that prohibits therapy treatments, dietary restrictions) will be excluded.
* Females who are pregnant will not be permitted in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of individuals that complied with treatment/intervention | up to 6 months
  Compliance among treatment group in meeting 2 g/kg protein goal as measured by protein tracking app and in protein supplements provided will be measured.
Percentage of frequency individuals successfully used the protein tracking app | up to 6 months
  Compliance in usage of protein tracking app will be recorded. The number of days they logged in and recorded their intake vs. total potential days to provide % value of diet protein compliance.
Percentage of physical therapy visits attended by individuals | up to 6 months
  Compliance in physical therapy will be recorded.
Percentage counseling sessions attended by individuals | up to 6 months
  Compliance in attending nutritional counseling sessions will be recorded.

SECONDARY OUTCOMES:
Single Leg Hop Test | baseline and up to 6 month
  Functional healing time based on single leg hop test. The distance the participant hopped on one leg will be recorded and measured in centimeters. This will be done three times and an average will be given.
Six Meter Timed Hop Test | baseline and up to 6 month
  Functional healing time based six meter timed hop test. The time it took the participant to hop six meters on foot will be measured and recorded.
Change in strength in leg flexion and extension | baseline and up to 6 month
  Strength in leg flexion and extension, as measured by Biodex machine
Change in muscle hypertrophy | baseline and up to 6 month
  depth of vastus medialis as measured at each nutritional advising appointment with counselor via ultrasound and thigh circumference.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Miller, Ph.D., Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available for health history, surgery type, clinical outcomes, and length of time in study.
Supporting Information: Study Protocol
Time Frame: The data will be available once the study is completed for a 12-month period.
Access Criteria: Interested parties should contact the PI- Gary Miller - for access

REFERENCES:
- [Background] Mather RC 3rd, Koenig L, Kocher MS, Dall TM, Gallo P, Scott DJ, Bach BR Jr, Spindler KP; MOON Knee Group. Societal and economic impact of anterior cruciate ligament tears. J Bone Joint Surg Am. 2013 Oct 2;95(19):1751-9. doi: 10.2106/JBJS.L.01705. PMID 24088967
- [Background] Ohura T, Nakajo T, Okada S, Omura K, Adachi K. Evaluation of effects of nutrition intervention on healing of pressure ulcers and nutritional states (randomized controlled trial). Wound Repair Regen. 2011 May-Jun;19(3):330-6. doi: 10.1111/j.1524-475X.2011.00691.x. PMID 21539650
- [Background] Iizaka S, Kaitani T, Nakagami G, Sugama J, Sanada H. Clinical validity of the estimated energy requirement and the average protein requirement for nutritional status change and wound healing in older patients with pressure ulcers: A multicenter prospective cohort study. Geriatr Gerontol Int. 2015 Nov;15(11):1201-9. doi: 10.1111/ggi.12420. Epub 2014 Dec 11. PMID 25496092
- [Background] Hurt RT, McClave SA, Martindale RG, Ochoa Gautier JB, Coss-Bu JA, Dickerson RN, Heyland DK, Hoffer LJ, Moore FA, Morris CR, Paddon-Jones D, Patel JJ, Phillips SM, Rugeles SJ, Sarav Md M, Weijs PJ, Wernerman J, Hamilton-Reeves J, McClain CJ, Taylor B. Summary Points and Consensus Recommendations From the International Protein Summit. Nutr Clin Pract. 2017 Apr;32(1_suppl):142S-151S. doi: 10.1177/0884533617693610. PMID 28388374
- [Background] Pasiakos SM, McLellan TM, Lieberman HR. The effects of protein supplements on muscle mass, strength, and aerobic and anaerobic power in healthy adults: a systematic review. Sports Med. 2015 Jan;45(1):111-31. doi: 10.1007/s40279-014-0242-2. PMID 25169440
- [Background] Cresci GA. Nutrition Support for the Critically Ill Patient: A Guide to Practice. Boca Raton, FL. CRC Press, 2005.
- [Background] Daly RM, O'Connell SL, Mundell NL, Grimes CA, Dunstan DW, Nowson CA. Protein-enriched diet, with the use of lean red meat, combined with progressive resistance training enhances lean tissue mass and muscle strength and reduces circulating IL-6 concentrations in elderly women: a cluster randomized controlled trial. Am J Clin Nutr. 2014 Apr;99(4):899-910. doi: 10.3945/ajcn.113.064154. Epub 2014 Jan 29. PMID 24477043
- [Background] Crickmer M, Dunne CP, O'Regan A, Coffey JC, Dunne SS. Benefits of post-operative oral protein supplementation in gastrointestinal surgery patients: A systematic review of clinical trials. World J Gastrointest Surg. 2016 Jul 27;8(7):521-32. doi: 10.4240/wjgs.v8.i7.521. PMID 27462395
- [Background] Fulgoni VL 3rd. Current protein intake in America: analysis of the National Health and Nutrition Examination Survey, 2003-2004. Am J Clin Nutr. 2008 May;87(5):1554S-1557S. doi: 10.1093/ajcn/87.5.1554S. PMID 18469286
- [Background] Campbell WW, Johnson CA, McCabe GP, Carnell NS. Dietary protein requirements of younger and older adults. Am J Clin Nutr. 2008 Nov;88(5):1322-9. doi: 10.3945/ajcn.2008.26072. PMID 18996869
- [Background] Antonio J, Ellerbroek A, Silver T, Vargas L, Tamayo A, Buehn R, Peacock CA. A High Protein Diet Has No Harmful Effects: A One-Year Crossover Study in Resistance-Trained Males. J Nutr Metab. 2016;2016:9104792. doi: 10.1155/2016/9104792. Epub 2016 Oct 11. PMID 27807480
- [Background] Naclerio F, Larumbe-Zabala E. Effects of Whey Protein Alone or as Part of a Multi-ingredient Formulation on Strength, Fat-Free Mass, or Lean Body Mass in Resistance-Trained Individuals: A Meta-analysis. Sports Med. 2016 Jan;46(1):125-137. doi: 10.1007/s40279-015-0403-y. PMID 26403469
- [Background] Fabre M, Hausswirth C, Tiollier E, Molle O, Louis J, Durguerian A, Neveux N, Bigard X. Effects of Postexercise Protein Intake on Muscle Mass and Strength During Resistance Training: Is There an Optimal Ratio Between Fast and Slow Proteins? Int J Sport Nutr Exerc Metab. 2017 Oct;27(5):448-457. doi: 10.1123/ijsnem.2016-0333. Epub 2017 Apr 19. PMID 28422532
- [Background] Alisson-Silva F, Kawanishi K, Varki A. Human risk of diseases associated with red meat intake: Analysis of current theories and proposed role for metabolic incorporation of a non-human sialic acid. Mol Aspects Med. 2016 Oct;51:16-30. doi: 10.1016/j.mam.2016.07.002. Epub 2016 Jul 12. PMID 27421909
- [Background] Schoenfeld BJ, Aragon A, Wilborn C, Urbina SL, Hayward SE, Krieger J. Pre- versus post-exercise protein intake has similar effects on muscular adaptations. PeerJ. 2017 Jan 3;5:e2825. doi: 10.7717/peerj.2825. eCollection 2017. PMID 28070459
- [Background] Trommelen J, van Loon LJ. Pre-Sleep Protein Ingestion to Improve the Skeletal Muscle Adaptive Response to Exercise Training. Nutrients. 2016 Nov 28;8(12):763. doi: 10.3390/nu8120763. PMID 27916799
- [Background] Coughlin SS, Whitehead M, Sheats JQ, Mastromonico J, Hardy D, Smith SA. Smartphone Applications for Promoting Healthy Diet and Nutrition: A Literature Review. Jacobs J Food Nutr. 2015;2(3):021. PMID 26819969
- [Background] Krebs P, Prochaska JO, Rossi JS. A meta-analysis of computer-tailored interventions for health behavior change. Prev Med. 2010 Sep-Oct;51(3-4):214-21. doi: 10.1016/j.ypmed.2010.06.004. Epub 2010 Jun 15. PMID 20558196
- [Background] Burke LE, Conroy MB, Sereika SM, Elci OU, Styn MA, Acharya SD, Sevick MA, Ewing LJ, Glanz K. The effect of electronic self-monitoring on weight loss and dietary intake: a randomized behavioral weight loss trial. Obesity (Silver Spring). 2011 Feb;19(2):338-44. doi: 10.1038/oby.2010.208. Epub 2010 Sep 16. PMID 20847736
- [Background] Harrison GG, Galal OM, Ibrahim N, Khorshid A, Stormer A, Leslie J, Saleh NT. Underreporting of food intake by dietary recall is not universal: a comparison of data from egyptian and american women. J Nutr. 2000 Aug;130(8):2049-54. doi: 10.1093/jn/130.8.2049. PMID 10917924
- [Background] Novotny JA, Rumpler WV, Riddick H, Hebert JR, Rhodes D, Judd JT, Baer DJ, McDowell M, Briefel R. Personality characteristics as predictors of underreporting of energy intake on 24-hour dietary recall interviews. J Am Diet Assoc. 2003 Sep;103(9):1146-51. doi: 10.1016/s0002-8223(03)00975-1. PMID 12963942
- [Background] Haynes RB, McDonald HP, Garg AX. Helping patients follow prescribed treatment: clinical applications. JAMA. 2002 Dec 11;288(22):2880-3. doi: 10.1001/jama.288.22.2880. PMID 12472330
- [Background] Naclerio F, Larumbe-Zabala E, Ashrafi N, Seijo M, Nielsen B, Allgrove J, Earnest CP. Effects of protein-carbohydrate supplementation on immunity and resistance training outcomes: a double-blind, randomized, controlled clinical trial. Eur J Appl Physiol. 2017 Feb;117(2):267-277. doi: 10.1007/s00421-016-3520-x. Epub 2016 Dec 27. PMID 28028619
- [Background] Askanazi J, Carpentier YA, Jeevanandam M, Michelsen CB, Elwyn DH, Kinney JM. Energy expenditure, nitrogen balance, and norepinephrine excretion after injury. Surgery. 1981 Apr;89(4):478-84. PMID 7209795
- [Background] Crane CW, Picou D, Smith R, Waterlow JC. Protein turnover in patients before and after elective orthopaedic operations. Br J Surg. 1977 Feb;64(2):129-33. doi: 10.1002/bjs.1800640212. PMID 890247
- [Background] Herzog MM, Marshall SW, Lund JL, Pate V, Mack CD, Spang JT. Incidence of Anterior Cruciate Ligament Reconstruction Among Adolescent Females in the United States, 2002 Through 2014. JAMA Pediatr. 2017 Aug 1;171(8):808-810. doi: 10.1001/jamapediatrics.2017.0740. PMID 28604937
- [Background] Millward DJ, Jackson AA. Protein/energy ratios of current diets in developed and developing countries compared with a safe protein/energy ratio: implications for recommended protein and amino acid intakes. Public Health Nutr. 2004 May;7(3):387-405. doi: 10.1079/PHN2003545. PMID 15153271
- [Background] Phillips SM. Current Concepts and Unresolved Questions in Dietary Protein Requirements and Supplements in Adults. Front Nutr. 2017 May 8;4:13. doi: 10.3389/fnut.2017.00013. eCollection 2017. PMID 28534027